CLINICAL TRIAL: NCT01972087
Title: Simulation Training to Improve 911 Dispatcher Identification of Cardiac Arrest
Acronym: STAT911
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Hendrika Meischke, Professor, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 44640-EJ; 5R18HS021658-02 (AHRQ)
Record Dates: First submitted 2013-10-18; First posted 2013-10-30 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participants randomized to the control arm receive no telephone simulation training.
- Simulation Training (Experimental): Participants randomized to the intervention arm receive telephone simulation training.
  Interventions: Behavioral: Telephone simulation training

INTERVENTIONS:
Behavioral: Telephone simulation training — The intervention consists of four 20-minute telephone simulation training sessions over a 4 month period (one session each month). Each 20-minute training session will include 3 simulated 9-1-1 calls, performed by a standardized caller (trained actor) and feedback will be provided right away by a trained observer who takes notes during the simulation calls and discusses the teaching points after the session. In total, the 9-1-1 dispatchers will receive 12 different simulated calls.
  Arms: Simulation Training

SUMMARY:
This study is to test the use of simulation training to improve 9-1-1 telecommunicators' call processing and response. Training sessions will expose 9-1-1 telecommunicators to several realistic emergency situations through mock 9-1-1 calls with a trained actor playing the part of a reporting party, followed immediately by feedback on call handling provided by a trained call observer. Investigators hypothesize that simulation followed by trained observer-directed feedback will increase correct triage of medical emergency and delivery of pre-arrival instructions during simulated calls and in actual 9-1-1 calls.

ELIGIBILITY:
Inclusion Criteria: 9-1-1 call-center call receivers. -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in elapsed seconds from call answer to start of telephone-cardiopulmonary resuscitation (T-CPR) instructions in cardiac arrest calls in simulations and in actual calls. | Once monthly over 4 months (during simulations); at event (actual cardiac arrest 9-1-1 call) over 12 months.

SECONDARY OUTCOMES:
Change in proportion of calls with querying behaviors compliant with the "all-callers" interviewing protocol. | Once monthly over 4 months (during simulations); at event (actual cardiac arrest 9-1-1 call) over 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hendrika Meischke, PhD, Principal Investigator — University of Washington

REFERENCES:
- [Derived] Stangenes SR, Painter IS, Rea TD, Meischke H. Delays in recognition of the need for telephone-assisted CPR due to caller descriptions of chief complaint. Resuscitation. 2020 Apr;149:82-86. doi: 10.1016/j.resuscitation.2020.02.013. Epub 2020 Feb 20. PMID 32088255
- [Derived] Meischke H, Painter IS, Stangenes SR, Weaver MR, Fahrenbruch CE, Rea T, Turner AM. Simulation training to improve 9-1-1 dispatcher identification of cardiac arrest: A randomized controlled trial. Resuscitation. 2017 Oct;119:21-26. doi: 10.1016/j.resuscitation.2017.07.025. Epub 2017 Jul 29. PMID 28760696
- [Derived] Meischke H, Painter I, Turner AM, Weaver MR, Fahrenbruch CE, Ike BR, Stangenes S. Protocol: simulation training to improve 9-1-1 dispatcher identification of cardiac arrest. BMC Emerg Med. 2016 Feb 1;16:9. doi: 10.1186/s12873-016-0073-6. PMID 26830676